CLINICAL TRIAL: NCT04464005
Title: Comparison Between Pads With Cold Solution of Magnesium Sulfate or Cold Water to Treat Pain and Improve Healing of the Perineum After Vaginal Delivery. A Prospective, Randomized, Double-blind Controlled Study.
Brief Title: Comparison Between Pads With Cold Solution of Magnesium Sulfate or Cold Water Postpartum Perineal Pain and Healing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 112-19
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-09

CONDITIONS: Women After Delivery With Perineal Pain
MeSH Terms: interventions — Magnesium Sulfate; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pads with cold magnesium sulfate 33% solution (Experimental)
  Interventions: Drug: Magnesium sulfate 33% solution
- Pads with cold water (Placebo Comparator)
  Interventions: Other: Cold water

INTERVENTIONS:
Drug: Magnesium sulfate 33% solution — Topical pads with cold magnesium sulfate 33% solution will be given 5 times/day for 15 minutes
  Arms: Pads with cold magnesium sulfate 33% solution
Other: Cold water — Topical pads with cold water will be given 5 times/day for 15 minutes
  Arms: Pads with cold water

SUMMARY:
Perineal pain after delivery is common and is caused by local bruising or episiotomy. The pain may last for several days or months. Thus, several analgesic methods are offered. Topical magnesium sulfate 33% solution is a common treatment for perineal pain, wound treatment and alleviation of swelling. Yet, the efficacy of this treatment was not tested sufficiently in a clinical trials.

In the present study we will compare the efficacy of topical magnesium sulfate versus cold water for perineal pain and improved perineal healing after delivery.

Women after vaginal delivery (spontaneous or operative) with pain score of 3 in 0-10 numeric rating scale (NRS) will randomly be allocated to receive either pad with cold magnesium sulfate 33% solution or cold water. Pain score and healing parameters will be assessed at baseline, after one day of treatment and after two days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Woman after spontaneous or operative vaginal delivery
* Perineal pain score of at least 2 NRS

Exclusion Criteria:

* Women after cesarean delivery
* Refuse to participate
* Under 18 years of age
* Magnesium sulfate treatment not related to the study
* Contraindication for magnesium sulfate treatment
* Workers of the local obstetric department

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of women with perineal pain score< 3 NRS at the day after treatment initiation | 24 hours post enrollment
Perineal pain intensity according to NRS scale at the day after treatment initiation | 24 hours post enrollment

SECONDARY OUTCOMES:
Degree of perineal healing using the REEDA scale | 2 days
Perineal pain intensity according to NRS scale two days after treatment initiation | 2 days (if still in hospital)
Rate of women with improvement in hemorrhoids characteristics in women with hemorrhoids | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Baruch Padeh Medical center, Poriya, Tiberias, North, Israel

IPD SHARING:
Plan to Share IPD: Undecided